CLINICAL TRIAL: NCT03242161
Title: Development of LabPatch-alcohol: A Wearable Biosensor for Detecting Alcohol in Interstitial Fluid
Brief Title: Development of LabPatch-alcohol as a Noninvasive Skin Patch to Detect Blood Alcohol Concentrations
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Director, McLean Imaging Center, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017P001502
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Intervention Model Description: All participants assigned to have a lab patch-alcohol applied to skin and then receive a single dose of alcohol and then the patch measures how much alcohol appears in interstitial fluid. This is compared to the blood alcohol concentrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LabPatch-alcohol (Experimental): All subjects will be administered alcohol and then monitored by a non-invasive alcohol sensor
  Interventions: Diagnostic Test: LabPatch-alcohol

INTERVENTIONS:
Diagnostic Test: LabPatch-alcohol — a wearable, non-invasive biosensor Band-Aid like patch that is designed to detect real-time changes in interstitial alcohol concentrations in human subjects after they have consumed alcohol

SUMMARY:
This study is designed to test LabPatch-alcohol, a wearable, non-invasive biosensor Band-Aid like patch that is designed to detect real-time changes in interstitial alcohol concentrations in human subjects. The changes in interstitial alcohol concentrations will be compared to blood alcohol concentrations to determine the patch's validity against the gold standard.

DETAILED DESCRIPTION:
Nanotechnology has the potential to become a powerful tool in addiction medicine. The potential utility for passive, non-invasive wearable alcohol monitors is great and could play a major role in public safety as well as in both research, clinical, and treatment settings. Clinitech, LLC has developed LabPatch, an electronic bandage that continuously and imperceptibly samples interstitial fluid from the skin surface and measures relevant biomarkers in the fluid. The patch uses novel nanowire technology to sample the interstitial fluid from just underneath the skin and then uses an electrochemical reaction to measure either glucose or alcohol concentration. The participants' interstitial alcohol concentration (IAC) will be measured via LabPatch-alcohol at the same time points as blood samples so that a direct comparison can be made. Thus, the LabPatch-alcohol will be tested as the participant's BAC rises and falls through the legally intoxicated concentration (0.08%), and the goal is to match measures obtained via the prototype LabPatch-alcohol with whole blood alcohol concentrations. The LabPatch operational circuit lies on the underside of the bandage. The circuit surface is placed in contact with the skin by the application of the elastic adhesive bandage with a contact tension that provides modest pressure, as in the case of a conventional wound bandage. The temperature of the skin is measured electrically and the consistency of temperature is used to verify good contact and to monitor continued contact. The entire process takes 3-5 seconds to collect the sample, a pause for 1 sec and then 3 additional seconds to conduct the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of understanding and complying with the protocol
* Good physical and mental health (normal physical exam, ECG, blood and urine chemistries, including absences of history or laboratory evidence of diabetes)
* Body Mass Index between 18-30, inclusive
* Age 21-50 years (age will be verified by driver's license or other valid form of identification)
* Have used alcohol, on average, between 5-15 drinks per week over the past 6 months.
* Have a stable living situation with current postal address

Exclusion Criteria:

* Meets criteria for current alcohol or substance use disorders (Past alcohol or substance use disorders greater than 3 years ago is acceptable)
* Concurrent diagnosis of Axis I disorder
* bMaintained on an antipsychotic or antidepressant medication; taking prescription medications except certain short-term anti-fungal agents and some tropical creams for dermal conditions
* Heavy alcohol drinkers (greater than 15 drinks per week)
* Tobacco use greater than 5 cigarettes per day
* History of major head trauma resulting in cognitive impairment or history of seizure disorder
* Heavy caffeine use (greater than 500 mg on a regular daily basis)
* Subject has active hepatitis and/or aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3x the upper limit of normal
* For female volunteers, a positive pregnancy test

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Interstitial and Blood Alcohol Concentrations | Both samples will be collected at baseline and at 2.5 to 5 minute intervals for up to 2.5 hrs after a 0.9 g/kg dose of alcohol.
  Interstitial (from the skin surface) alcohol concentrations will be obtained via the LabPatch band-aid while at the same time blood samples will be collected in an attempt to correlate the two. The LabPatch-alcohol is a completely noninvasive device and the goal is to determine is precision against the gold standard--blood alcohol concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Lukas, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No